CLINICAL TRIAL: NCT07209943
Title: Cognixion Pass Through Study
Brief Title: Augmented Reality BCI Longitudinal Study for Persons With ALS, Stroke, TBI and SCI Utilizing Cognixion + Apple Vision Pro
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cognixion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: COG-AVP-002
Record Dates: First submitted 2025-09-18; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis); TBI Traumatic Brain Injury; SCI - Spinal Cord Injury; Stroke
Keywords: usability study; augmented reality; brain computer interface; als; generative AI; agentic; spinal cord injury; traumatic brain injury
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Brain Injuries, Traumatic; Spinal Cord Injuries; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Usability Study (Experimental): Participants will utilize the Cognixion + Apple Vision Pro device and associated communication and computer control software for practice and communication tasks as prescribed by the study administrator. Various modalities, including pure BCI and ET-BCI will be available to users.
  Interventions: Device: Cognixion + Apple Vision Pro

INTERVENTIONS:
Device: Cognixion + Apple Vision Pro — An Apple Vision Pro device, integrated with Cognixion's brain sensing band and Assisted Reality software. The integrated device enables users to construct AI assisted communication and computer control commands using a combination of attention, eye gaze and head pose.

SUMMARY:
The goal of this study is refine the usability of a BCI capable communication platform.

The study will take place in the United States area and will enroll up to 10 participants with late stage ALS, traumatic brain injury (TBI) or spinal cord injury (SCI) that have assistive communication and computer control needs. Each subject will receive an integrated Cognixion + Apple Vision Pro device that includes an augmented reality brain computer interface and associated communication software. The study duration is 3-4 months for each participant.

The key questions that will be addressed in this study are:

1. Identify the ability of individuals with target indications to use the integrated Cognixion-Apple Vision Pro system to communicate effectively.
2. Identify the ability of such individuals to learn to use BCI, ET-BCI and other modalities, and to measure their progress over time.
3. Identify the effectiveness of the different forms of input supported by the combined Cognixion-Apple Vision Pro system (BCI, eye-tracking) in allowing such individuals to communicate and have agency.
4. Identify how input such as BCI can be optimized to suit the needs of individuals (e.g., specific frequencies that work best for an individual, SNR with different frequencies, number of targets, length of recording for each frequency) and improve overall usability.
5. Identify the extent to which personalization through a large language model (LLM) affects communication.
6. Identify the appropriate capabilities to enable through an agentic communication interface.

Key measures include:

ITR - information transfer rate SUS - system usability scale

ELIGIBILITY:
Inclusion criteria:

* Must have a designated on-site support individual who can be trained on the Cognixion system
* Fluent in understanding English
* 18 years or older
* Must have one of ALS, spinal cord injury or chronic brain injury and need an assistive communication device
* Must be able to engage in volitional eye opening and sustain eye opening independently for at least 30 minutes.
* Must have a way to communicate apart from using the Cognixion device such as vocalizations, head nod, eye blinks, eyebrow raises, etc. At a minimum, reliable, independent way of communicating "Yes" and "No"

Exclusion criteria:

* Disruption in English comprehension, either due to lack of fluent proficiency or due to a developmental/acquired language disorder (e.g. aphasia)
* Severely hearing impaired or deaf
* Sensitivity to flashing lights
* Claustrophobia related to the Apple Vision Pro with comfort adapter
* History of epilepsy and/or seizures
* Vision disorders restricting the visual field such as glaucoma, diplopia (double vision), nystagmus (involuntary eye movements)
* History of vertigo or other vestibular disorders
* Scalp that is prone to irritation, inflammation, injury, or infectious process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-16 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
System Usabilty Score | 3-4 months
  A score ranging from 0 to 100 that captures the usability the device and enables it to be compared with other human machine interface devices. This is an intrisic property of the device interface (hardware/software) and is not a healh outcome measure.
Information Transfer Rate (ITR) | 3-4 months
  The rate, in bits per minute, of information transfer for each of the device modalities. ITR is measured using a standardized selection procedure and is a measure the captures how efficient the device interface is. It is an essential measure of device throughput and is not related to any health outcome.

SECONDARY OUTCOMES:
Phrases per Minute | 3-4 months from training
  PPM is the number of complete phrases or compute rcommands that the user can construct in 1 minute. This is a usage metric that captures the efficiency of the device in predicting user utterances and does not relate to any health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Ullrich, Principal Investigator — Cognixion
Locations (1):
- Cognixion HQ, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Usability insights related to this use case on this type of device will be shared with other accessibility and BCI researchers at conference events and through publications. This data will be anonymized prior to sharing.
Supporting Information: CSR
Time Frame: Clinical study report will be shared upon request once complete. Estimated to occur no sooner than April 1 2026.
Access Criteria: Anonymized clinical study report will be made available to clinical researchers, upon request and validation.

REFERENCES:
- [Background] Wolpaw JR, Bedlack RS, Reda DJ, Ringer RJ, Banks PG, Vaughan TM, Heckman SM, McCane LM, Carmack CS, Winden S, McFarland DJ, Sellers EW, Shi H, Paine T, Higgins DS, Lo AC, Patwa HS, Hill KJ, Huang GD, Ruff RL. Independent home use of a brain-computer interface by people with amyotrophic lateral sclerosis. Neurology. 2018 Jul 17;91(3):e258-e267. doi: 10.1212/WNL.0000000000005812. Epub 2018 Jun 27. PMID 29950436
- [Background] Kellmeyer P, Grosse-Wentrup M, Schulze-Bonhage A, Ziemann U, Ball T. Electrophysiological correlates of neurodegeneration in motor and non-motor brain regions in amyotrophic lateral sclerosis-implications for brain-computer interfacing. J Neural Eng. 2018 Aug;15(4):041003. doi: 10.1088/1741-2552/aabfa5. Epub 2018 Apr 20. PMID 29676287
- [Background] Lewis, J. R. (2018). The System Usability Scale: Past, Present, and Future. International Journal of Human-Computer Interaction, 34(7), 577-590